CLINICAL TRIAL: NCT00285675
Title: A Continuation Study of DN-101 (Calcitriol) and Docetaxel in Subjects Previously Enrolled in Studies DN101-002 or DN101-004
Brief Title: Study of DN-101 (Calcitriol) and Docetaxel in Subjects Previously Enrolled in Studies DN101-002 or DN101-004
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Novacea (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 011-016
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2006-05-31 (Estimated); Status verified 2006-01

CONDITIONS: Androgen Independent Prostate Cancer (AIPC); Non Small Cell Lung Cancer (NSCLC)
Keywords: Calcitriol, DN-101, Androgen Independent Prostate Cancer (AIPC), Prostate Cancer, Non Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms | interventions — Calcitriol; Pharmaceutical Preparations

INTERVENTIONS:
Drug: DN-101 (calcitriol) - Drug

SUMMARY:
The purpose of this study is to monitor the safety of continued DN-101 and docetaxel treatment for subjects previously enrolled in DN101-002 (ASCENT) or DN101-004 (NSCLC) Studies.

DETAILED DESCRIPTION:
This is a multicenter, open-label trial of DN-101 and docetaxel combination therapy to monitor the safety of ongoing DN-101 and docetaxel treatment for subjects previously enrolled in DN101-002 or DN101-004 studies. For subjects enrolled in DN101-002 study, only subjects randomized to the DN-101 treatment arm and are currently receiving study drug (including subjects on study suspension / holiday) will be included in the current study. For subjects enrolled in DN101-004 study, only subjects who are receiving study treatment will be included.

Safety will be assessed throughout the study. Safety evaluations will consist of a modified physical exam (vital signs and weight) and laboratory assessments. Modified physical exam should be performed at the beginning of each treatment cycle. Docetaxel-related laboratory assessments will be performed per standard of care as noted in the labeling. DN-101-related laboratory assessments for serum calcium and serum creatinine will be performed at the beginning of each treatment cycle. Clinically significant abnormal laboratory values will be reported as adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in DN101-002 or DN101-004 studies, where the subject received at least one dose of DN-101
* Able and willing to give written informed consent

Exclusion Criteria:

* Disease progression or unacceptable toxicity while previously enrolled in DN101-002 or DN101-004 studies
* Prior investigational therapy other than DN-101 within 30 days of enrollment
* Known hypersensitivity to calcitriol
* Pregnancy (women of childbearing potential only)
* Greater than 90 days has elapsed from termination of DN101-002 or DN101-004 studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2006-04; Study Completion 2008-01

CONTACTS AND LOCATIONS:
Locations (13):
- United States (11):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Kaiser Permanente Medical Group, Northern California, Vallejo, California
  - Columbia Presbyterian Medical Center, New York, New York
  - Piedmont Hematology Oncology Associates, Winston-Salem, North Carolina
  - NW Kaiser Permanente Portland, Portland, Oregon
  - Alta Bates Comprehensive Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh,William Copper Ambulatory Care, Pavillion Hellman Cancer Center, Pittsburgh, Pennsylvania
  - Tyler Cancer Center, Tyler, Texas
  - Northwest Cancer Specialists Vancouver Office, Vancouver, Washington
- Canada (2):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Department of Medicine, Edmonton, Alberta